CLINICAL TRIAL: NCT05522868
Title: An Open-label, Multicenter, Phase 1 Clinical Trial to Evaluate MTD, Safety, PK/PD and Preliminary Anti-tumor Activity of SB17170 in Patients With Locally Advanced or Metastatic Solid Tumors Who Have Failed Standard of Care
Brief Title: SB17170 Phase 1 Clinical Trial in Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SPARK Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SMARTT-001
Record Dates: First submitted 2022-08-25; First posted 2022-08-31 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor

STUDY DESIGN:
Intervention Model Description: Traditional 3+3 Dose Ascending design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Other): SB17170 initial dose: 300 mg/d per day, 3 to 6 subjects per cohort
  Interventions: Drug: SB17170
- Cohort 2 (Other): SB17170 dose: 600 mg/d per day, 3 to 6 subjects per cohort
  Interventions: Drug: SB17170
- Cohort 3 (Other): SB17170 dose: 1000 mg/d per day, 3 to 6 subjects per cohort
  Interventions: Drug: SB17170

INTERVENTIONS:
Drug: SB17170 — SB17170 capsules, Oral administration 21days/cycle

SUMMARY:
Phase 1 Open-label, multicenter, dose escalation, dose expansion study

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase 1 clinical trial to evaluate the maximum tolerated dose, safety, pharmacokinetic/pharmacodynamic characteristics and preliminary anti-tumor activity of SB17170 when administered alone(1a) and co-administered with standard of care(1b) to patients with locally advanced or metastatic solid tumors who have failed standard of care.

1 cycle of treatment of this clinical trial is 21 days, and tumors are assessed every 2 cycles.

ELIGIBILITY:
Inclusion Criteria:

* A patient with a histologically or cytologically confirmed diagnosis of locally advanced or metastatic solid tumors.
* A person who has failed the known standard of care or has developed resistance to the standard of care and no longer has applicable standard of care
* A patient with at least one measurable lesion according to the RECIST v1.1 criteria.
* A person with Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1.
* Those with an expected survival period of 3 months or more at the discretion of of the investigator.

Exclusion Criteria:

* A patient who has received drugs targeting High Mobility Group Box 1 (HMGB1).
* A patient who has received or is undergoing chemotherapy (including chemotherapy, radiation therapy, immunotherapy, hormone therapy, targeted therapy, biological products, and tumor embolization) within 28 days from the first administration date of the investigational drug.
* A person who needs to take contraindicated drugs or is expected to take them during the study period.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of SB17170 | At the end of Cycle 1 (each cycle is 21 days)
  Evaluate DLT to estimate the maximum tolerated dose (MTD), and determine a recommended Phase 2 dose (RP2D).

SECONDARY OUTCOMES:
Pharmacokinetic(Cmax) | At Day1 and D21 of Cycle 1 (each cycle is 21 days)
  Peak Plasma Concentration
Pharmacokinetic(Tmax) | At Day1 and D21 of Cycle 1 (each cycle is 21 days)
  Time to Peak Plasma Concentration
Pharmacokinetic(AUC) | At Day1 and D21 of Cycle 1 (each cycle is 21 days)
  Area under the plasma concentration versus time curve
The anti-tumor activity with RECIST v1.1 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, up to 100weeks
  CT/MRI every 6 weeks
Pharmacodynamics(TIL) | At Day1 and D22 of Cycle 1 (each cycle is 21 days)
  Tumor infiltrated lymphocyte in Tumor tissue
Pharmacodynamics(TAM) | At Day1 and D21 of Cycle 1 (each cycle is 21 days)
  Tumor Associated Macrophage at Tumor Tissue
Pharmacodynamics(T cell activation) | At Day1 and D21 of Cycle 1 and D1 of each cycle (each cycle is 21 days)
  T cell activation in Blood
Pharmacodynamics(PD-L1) | At Day1 and D21 of Cycle 1 and D1 of each cycle (each cycle is 21 days)
  PD-L1 in Blood and D1 of each cycle
Pharmacodynamics(High Mobility Group Box 1 ) | At Day1 and D21 of Cycle 1 and D1 of each cycle (each cycle is 21 days)
  HMGB1 in Blood and Tissue
Pharmacodynamics(S100A8) | At Day1 and D21 of Cycle 1 t and D1 of each cycle (each cycle is 21 days)
  S100A8 in Blood
Pharmacodynamics(S100A9) | At Day1 and D21 of Cycle 1 and D1 of each cycle(each cycle is 21 days)
  S100A9 in Blood
Pharmacodynamics(CXCL8) | At Day1 and D21 of Cycle 1 and D1 of each cycle(each cycle is 21 days)
  CXCL8 in Blood
Pharmacodynamics(MDSC) | At Day1 and D21 of Cycle 1 and D1 of each cycle(each cycle is 21 days)
  Rate of Myeloid-Drived Suppressor Cell in Blood

CONTACTS AND LOCATIONS:
Overall Officials: Soojin Jun, Study Director — SPARK Biopharma
Locations (3):
- South Korea (3):
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No